CLINICAL TRIAL: NCT02152722
Title: Breath Test for Biomarkers in Humans Receiving Total Body Irradiation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Menssana Research, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Memorial Sloan Kettering Cancer Center (Other); Emory University (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: MR 2012 TBI
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Radiation Injury
Keywords: Breath test; Volatile Organic Compounds; VOC; oxidative stress; radiation biodosimetry; metabolomics; GCxGC TOF-MS
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Body Irradiation Subjects: Subjects undergoing total body irradiation prior to chemotherapy. It is expected that all of these subjects will be receiving ablative radiation prior to bone marrow transplant. Breath will be collected before and after the first radiation exposure on each day of total body irradiation.

SUMMARY:
The effect of radiation on normal tissue varies widely between individuals. Consequently, a test to measure tissue response to radiation could be clinically useful by permitting more accurate titration of dosage in patients undergoing radiotherapy. Also, in view of emerging concerns about possible nuclear terrorism a test for exposure to radiation might also be useful in evaluating victims of a "dirty bomb" explosion. A number of different techniques have been previously reported in epidemiological studies for the estimation of prior radiation exposure. This study explores one approach to estimating radiation exposure by measurement of increased oxidative stress which can be detected by a breath test.

In this study subjects undergoing significant exposure to therapeutic radiation will provide breath samples for analysis in a central laboratory. The hypothesis of the study is that the analysis of these samples will lead to the identification of a set of markers of radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Subject is willing and able to cooperate with study and give signed informed consent to participate
3. Subject has been diagnosed with a condition that requires treatment with a TBI protocol of daily irradiation for one to five days
4. Actively smoking subjects, as well as never smokers and former smokers are eligible for the study so long as a complete smoking consumption history can be recorded
5. Subject will be available for follow-up breath tests following each session of TBI. Subjects receiving only one day of TBI will be available for a follow-up 24-36 hours following TBI
6. Subject is an in-patient at the hospital

Exclusion Criteria:

1. Subject has had chemotherapy within preceding 21 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing total body irradiation prior to chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Radiation volatile organic compound (VOC) score | Each day of radiation exposure at time points between 1 day and 7 days post exposure.
  An algorithm for scoring the radiation exposure based on analysis of breath samples will be developed and applied to each breath sample collected. The hypothesis is that the scores will indicate radiation exposure, specifically exposure to more than 2 Gray at time points between 1 day and 7 days post exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, M.D., Principal Investigator — Menssana Research, Inc.
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Background] Phillips M, Byrnes R, Cataneo RN, Chaturvedi A, Kaplan PD, Libardoni M, Mehta V, Mundada M, Patel U, Ramakrishna N, Schiff PB, Zhang X. Detection of volatile biomarkers of therapeutic radiation in breath. J Breath Res. 2013 Sep;7(3):036002. doi: 10.1088/1752-7155/7/3/036002. Epub 2013 Jun 24. PMID 23793046